CLINICAL TRIAL: NCT01771302
Title: Randomized Clinical Trial on the Efficiency of PRGF-Endoret in Combination With a Bone Graft in Lateral Sinus Floor Elevation
Brief Title: Efficiency of PRGF-Endoret in Combination With a Bone Graft in Lateral Sinus Floor Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Collaborators: Biotechnology Institute IMASD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTI-EC/12/Biomat
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2015-07

CONDITIONS: Sinus Floor Augmentation
Keywords: PRGF-Endoret; Bone graft; Maxillary sinus; Vertical bone augmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bio-Oss (Active Comparator): the xenograft is of bovine origin where the organic phase has been eliminated.
  Interventions: Device: Bio-Oss
- calcium phosphate ceramic (Experimental): is a calcium phosphate biomaterial
  Interventions: Device: calcium phosphate ceramic

INTERVENTIONS:
Device: Bio-Oss — It is a bone substitute of bovine origin
  Arms: Bio-Oss
Device: calcium phosphate ceramic — It is a synthetic bone substitute ceramic that is composed of calcium and phosphate ions and prepared at high temperature
  Arms: calcium phosphate ceramic

SUMMARY:
This randomized clinical study investigates the efficiency of plasma rich in growth factors (PRGF-Endoret) in combination with bone grafts in the healing of bone and soft tissues after the performance of lateral sinus floor elevation.

The hypothesis of this study is that the use of PRGF-Endoret will produce similar bone formation regardless the type of bone graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients requiring implant prostheses oral rehabilitation.
* Patients with insufficient residual height in posterior maxilla requiring a sinus lift procedure to insert the implants

Exclusion Criteria:

* Not having complete the informed consent form.
* Sinusitis.
* Alcoholism.
* Suffering severe haematological disorder or disease.
* Be undergoing or having received radiotherapy, chemotherapy or immunosuppressive therapy, corticosteroids and / or anticoagulants, 30 days prior to the study inclusion.
* In usual treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or other anti-inflammatory drugs.
* Background of chronic hepatitis or liver cirrhosis.
* Diabetes mellitus with poor metabolic control (glycosylated hemoglobin above 9%)
* Patients undergoing dialysis.
* Presence of malignant tumors, hemangiomas or angiomas in the extraction area.
* History of ischemic heart disease in the last year.
* Pregnancy or intention to become pregnant during the study follow-up period.
* Metabolic bone disease
* Patients taking bisphosphonates drugs both orally and intravenously.
* In general, any inability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percentage of newly-formed bone | 6 months after surgical intervention
  The histomorphometrical analysis of the biopsies taken after 6 months of surgical intervention (time for dental implants insertion) will be performed to calculate the primary outcome

SECONDARY OUTCOMES:
Bone density | at baseline and after 6 months of intervention
  This data will be measured on the cone-beam CT scanners obtained at baseline and after 6 months of healing
Insertion torque | 6 months after surgical intervention
  At the time of implant insertion and initial insertion torque will be registered
Percentage of residual graft | 6 months after surgical intervention
  The histological analysis will determine the percentage of residual graft after 6 months of surgery.
Pain index | 7 days, 15 days, 1 month, 2 months, 6 months and 12 months after surgical intervention
  This will evaluate the intensity of pain the patient suffered due to the surgical intervention.
Healing index | 7 days, 15 days and 1 month after surgical intervention
  This index will evaluate the soft tissue healing.
Infection | 7 days, 15 days, 1 month, 2 months, 6 months and 12 months after surgical intervention
  Notify the infection of the graft material

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Anitua, MD, DDS, PhD, Principal Investigator — Clinica Eduardo Anitua
Locations (1):
- Clinica Eduardo Anitua, Vitoria-Gasteiz, Spain